CLINICAL TRIAL: NCT00209989
Title: Phase I/II Trial to Assess the Radiosensitizing Effect of ZARNESTRA in Patients With Glioblastoma Multiforme
Brief Title: Phase II Trial to Assess the Radiosensitizing Effect of ZARNESTRA in Patients With Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02 TETE 02
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma Multiforme; Zarnestra; Radiation therapy
MeSH Terms: conditions — Glioblastoma | interventions — tipifarnib

INTERVENTIONS:
Drug: Zarnestra — ZARNESTRA 100 bid (phase II recommended dose defined in phase I)will be administered continuously from one week prior to start of radiation therapy until the last day of radiation therapy.
Procedure: standard Radiation therapy — Radiotherapy will be focused on the initial tumour volume with a reasonable margin of safety (2 cm). A total dose of 60 Gray (Gy) will be given to the Clinical Target Volume

SUMMARY:
The purpose of this study is to determine the efficacy by the determination of the Time To Progression (TTP) in patients with resectable GBM or non surgical GBM with a size less than 5 cm treated with the combination of ZARNESTRA plus Radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed (histology or cytology), resectable or non resectable, glioblastoma multiforme with a size < 5 cm on MRI if non resectable
* Patients must be at least 7 days but no more than 2 months since surgery or biopsy.
* Patients must have an ECOG Performance Status ≤ 2.
* Patients must be aged 18
* Patient has signed the informed consent form

Exclusion Criteria:

* Patients with unresectable glioblastoma with a size >5 cm on MRI
* Patients with clinically apparent leptomeningeal metastases
* Patients with uncontrolled seizures despite standard anticonvulsant therapy
* Any prior systemic treatment (chemotherapy, immunotherapy, hormonal therapy) for glioblastoma multiforme
* Significantly abnormal haematological status as judged by:

Absolute neutrophil count (ANC) < 1500/mm3 (1.5*109/l) Platelet count <100,000/mm3 (100*109/l)

* Serum bilirubin >2 mg/dl (>34 mmol/l) or Transaminase >2.5x the upper limit of institutional normal or Creatinine >1.5 mg/dl (>132 mmol/l)
* Inability to co-operate with the treatment protocol
* Patients who cannot undergo imaging evaluations
* Participation in an investigational drug trial in the 30 days prior to selection
* Pregnant or nursing mothers. (Female patients of childbearing potential must use adequate contraception.)
* Any malignancy within the past five years. Exceptions are: superficial basal cell carcinoma or non-metastatic squamous cell cancer of the skin, cervix cancer (cervical intra-epithelial neoplasia -CIN or FIGO stage 1) or prostate intra-epithelial neoplasia (PIN), biochemical relapse free for at least 3 years.
* Any prior systemic chemotherapy in the past five years for any malignancy in the medical history
* Any concurrent disease that in the opinion of the investigator would constitute a hazard for participating in this study
* Known sensitivity to imidazole derivatives
* Patients under law protection
* Medical history of phlebitis or pulmonary embolism, thrombocytosis, myocardiopathy, or other relevant cardiac pathology (auricular flutter, auricular fibrillation)
* Medical history of immuno-allergic pneumopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Efficacy will be assessed by the determination of the Time To Progression (TTP) in patients with resectable GBM or non surgical GBM with a size less than 5 cm treated with the combination of ZARNESTRA plus Radiation therapy | time of study

SECONDARY OUTCOMES:
Objective response rate (RECIST and volumetric criteria) | time of study
Median survival, 6 month and 1 year survival rates | 6 month and 1 year
Safety of combination therapy of ZARNESTRA and RT, based on laboratory and clinical parameters | time of study

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth MOYAL, Dr, Principal Investigator — Institut Claudius Regaud
Locations (2):
- France (2):
  - Centre Jean Perrin, Clermont-Ferrand
  - Institut Claudius Regaud, Toulouse